CLINICAL TRIAL: NCT01229878
Title: Vitamin D Supplementation on Physical and Cognitive Function-Pilot Study
Brief Title: Vitamin D Supplementation in Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F7539-P
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Renal Dialysis; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Active Comparator): Hemodialysis Patients randomized to take Vitamin D supplements
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D)
- Placebo (Placebo Comparator): Hemodialysis Patients randomized to take placebo pills
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vitamin D) — 50,000 units of cholecalciferol or a placebo pill administered once a week for 6 months

SUMMARY:
This is a double-blind placebo controlled pilot study to determine if vitamin D supplementation in hemodialysis (HD) patients will improve physical function and cognition. HD patients have a high prevalence of vitamin D deficiency, cognitive impairment, and physical impairment. Despite standard clinical care with active IV vitamin D during dialysis, HD patients still have markedly low levels of nutritional or dietary vitamin D. IV treatment with vitamin D during dialysis is aimed at treating HD related bone disease. Recent literature shows that oral or nutritional vitamin D has multiple extra-skeletal effects including improvement in cognition and physical function. In this study, the investigators plan to administer oral vitamin D to vitamin D deficient HD patients already receiving standard care with IV vitamin D therapy. Patients will be randomized to receive either placebo or 50,000 IU of vitamin D (cholecalciferol) weekly for 6 months. The investigators' specific aims are to 1) Assess the benefits of correcting nutritional vitamin D deficiency on cognitive and physical function in HD patients receiving routine standard of care, 2) Assess the feasibility of recruiting HD patients for this study, and 3) Evaluate the proposed regimen for safely and effectively increasing nutritional vitamin D levels with oral supplementation. The investigators anticipate that correction of nutritional vitamin D deficiency to optimal levels will improve the high prevalence of cognitive impairment and physical impairment in this population. These results will be used as evidence to support a larger study aimed at treating nutritional vitamin D deficiency in all patients receiving HD. These results may also contribute to a change in current guidelines which place little emphasis on the monitoring and treatment of nutritional vitamin D levels in HD patients. These results are important for the Veteran dialysis population since many of them are required to perform high-level cognitive tasks such as management of complex medical regimens and physical tasks such as orchestrating independent transportation to and from HD sessions and multiple physician appointments.

DETAILED DESCRIPTION:
Patients will first be identified based on the inclusion criteria, then informed about the study and consented. Those who meet the exclusion criteria will be randomized to treatment or placebo. Enrolled participants will be randomized 2:1 to receive vitamin D (n=20) or placebo (n=10) for 6 months. All participants will be tested twice over two weeks to establish baseline values. Following baseline testing, the treatment group will receive 50,000 IU (standard replacement therapy) of oral cholecalciferol or placebo. The initial dose of cholecalciferol will be 50,000 IU weekly for 6 weeks. Vitamin D levels will then be measured. Participants who still have Vitamin D insufficiency ( 35 ng/ml) will remain on 50,000 IU of cholecalciferol for another 6 weeks, at which point Vitamin D levels will be measured again. Participants who reach 25-OH levels > 35 ng/ml will have their dosing regimen lessened to 10,000 IU weekly (maintenance dose) for the remainder of the 6 months. Participants receiving placebo will start taking the placebo maintenance dose after the first 6 weeks. For safety monitoring, 25(OH) vitamin D3 levels will also be re-measured at monthly intervals and followed by an independent medical monitor. In patients who have serum vitamin D levels 60ng/ml, the frequency of administration will be reduced to once a month. The participants will receive supplementation for a total of 6 months. At this time, vitamin D levels will be reassessed and participants will undergo follow-up functional assessments, and cognitive and immune testing.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HD for at least two weeks
* Receiving IV vitamin D supplementation according to National Kidney Foundation guidelines.
* Male or female with an between the ages of 45-89 years
* Veteran outpatient or stable community living center patient
* Able to ambulate independently or with an assistive device for at least 20 feet

Exclusion Criteria:

* 25-OH vitamin D level < 25 ng/ml
* Hypercalcemia
* Active malignancy within 6 months
* Receiving intravenous antibiotics for infection
* History of Dementia
* Hemoglobin < 8.5g
* History of conditions that interfere with postural instability (e.g. cerebellar disease, vestibular disease or any others that may present)
* Poor compliance with dialysis treatments (history of skipping 2 treatments per month for > 2 months)

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Post, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Hemodialysis Patients randomized to take Vitamin D supplements
  Cholecalciferol (Vitamin D): 50,000 units of cholecalciferol administered once a week for 6 months
- Placebo: Hemodialysis Patients randomized to take placebo pills
  Matching placebo pill administered once a week for 6 months
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 13 | 7
Completed | 10 | 6
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Hemodialysis Patients randomized to take placebo pills
  Placebo pill administered once a week for 6 months
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Hip Flexor Strength
Description: Neuromuscular Function - strength testing of hip flexors. Hip flexor strength measured using a push-pull muscle strength dynamometer. Participants performed a hip flexor exercise 3 times at each visit. The final result at each time point was an average of the 3 tries. Outcome measure is change between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 10 | 6
percent change | 20.34 (34.29) | 6.83 (36.44)

2. Secondary Outcome: Quality-of-Life Self Assessment
Description: questionnaire of physical/medical health
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Neuropsychological Assessments
Description: battery of neurocognitive tests
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Immune Function Assessments
Description: assay of immunity markers
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6.5 months - from the time of consent through the 6-month final visit.
Description: Arms/groups are combined for adverse event reporting due to the fluctuation of the vitamin D dosing regime. The dosing regime was adjusted from 50,000 IU to 10,000 IU of vitamin D depending on the participant's measured vitamin D level. If a participant's measured vitamin D level was greater than or equal to 60 ng/ml, the frequency of study drug administration was reduced to once a month instead of once a week. Each participant's timeline for dose adjustment is different.
Groups:
- Vitamin D: Hemodialysis Patients randomized to take Vitamin D supplements
  Cholecalciferol (Vitamin D): 50,000 units of cholecalciferol once a week for 6 months
Arm/Group | Vitamin D | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/13 | 1/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=13) | Placebo (N=7)
Hospitalization (Surgical and medical procedures) | 3 (3) | 0 (0)
ER visit (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
Prolonged Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Unstoppable bleeding from dialysis access port

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT01229878/Prot_SAP_000.pdf